CLINICAL TRIAL: NCT04197830
Title: Evaluation of Acute Post-thrombectomy Complications for Stroke
Acronym: Stroke ICU
Status: Completed | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Pierre Goffin, Principal Investigator, University of Liege
Other Study IDs: 00014
Record Dates: First submitted 2019-12-09; First posted 2019-12-13 (Actual); Last update posted 2020-11-13 (Actual); Status verified 2020-11

CONDITIONS: Stroke, Complication; Stroke, Acute; Stroke Hemorrhagic
MeSH Terms: conditions — Stroke; Hemorrhagic Stroke | interventions — Thrombectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Thrombectomy for stroke — Patients who have had thrombectomy for acute stroke.

SUMMARY:
Retrospective study to assess the incidence of acute complications after thrombectomy for stoke.

DETAILED DESCRIPTION:
Research in the computerized medical file of patients admitted to intensive care unit (ICU) in the last 5 years for a stroke.

Searching for acute complications during the ICU stay. Looking for hemorrhagic, acute renal failure, hemodynamic support, neurologic degradation.

ELIGIBILITY:
Inclusion Criteria:

* >18 year old
* ICU admitted patient for stroke and received thrombectomy

Exclusion Criteria:

* missing data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Retrospective cohort based on a computer medical record.
Sampling Method: Non-Probability Sample
Enrollment: 361 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Survival | day 0 to day 5
  death during ICU stay
hemorrhagic complication | day 1
  hemorrhagic complication base on CT scan at day 1
Neurological evaluation | day 0 to day 5
  Neurological evaluation based on Glasgow coma scale (from 3 pejorative to 15/15 good)
Evolution of renal function | day 0 to day 5
  Evaluation based on biological analyses : creatinine value based on daily routine blood analysis (in mg/dL).

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Goffin, MD, MSc, Principal Investigator — MontLegia Hospital, Groupe Santé CHC, Liège, Belgium
Locations (1):
- MontLegia Hospital, Liège, Belgium

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.